CLINICAL TRIAL: NCT03413631
Title: A Prenatal Mentalization-focused 4D Ultrasound and a Pregnancy Diary Intervention for Substance-abusing Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Foundation for Paediatric Research, Finland (Other); Academy of Finland (Other); Hospital District of Southwestern Finland (Other); University of Turku (Other)
Responsible Party: Principal Investigator, Eeva Ekholm, Consultant, MD, PhD, Docent, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13924
Record Dates: First submitted 2018-01-02; First posted 2018-01-29 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Substance-Related Disorders; Pregnancy, High Risk; Prenatal Care; Maternal-Fetal Relations; Parenting; Depression; Anxiety; Perinatal Outcome; Fetal Exposure During Pregnancy
Keywords: prenatal substance abuse; mentalization; prenatal depression; prenatal anxiety; maternal-fetal attachment; prenatal intervention; ultrasound; perinatal outcome; fetal exposure; parenting; parenthood; prenatal treatment
MeSH Terms: conditions — Substance-Related Disorders; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The participants were randomized into the intervention and control groups using a computer-generated block-randomization with block size of four. A separate randomisation assignment was used for women medication-assisted treatment for opioid addiction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prenatal mentalization intervention (Experimental): The intervention group participants were offered three mentalization-focused 4D interactive ultrasounds at 24, 30 and 34 gestational weeks and a mentalization-focused week-by-week pregnancy diary combined with three prenatal sessions and option for one session after delivery in addition to obstetric care as usual (see Prenatal obstetric treatment as usual).
  Interventions: Behavioral: Prenatal mentalization intervention; Other: Prenatal obstetric treatment as usual
- Prenatal obstetric treatment as usual (Active Comparator): The control group received obstetric care as usual in a tertiary setting. The comprehensive treatment as usual was conducted at the hospital antenatal outpatient clinic, including regular obstetric ultrasounds. The multidisciplinary treatment team, consisting of an obstetrician, a midwife, a social worker and a psychiatric nurse, assess and support health and psychosocial situation of the pregnant woman. The pregnant woman was referred to addiction and psychiatric treatment when needed.
  Interventions: Other: Prenatal obstetric treatment as usual

INTERVENTIONS:
Behavioral: Prenatal mentalization intervention
  Arms: Prenatal mentalization intervention
Other: Prenatal obstetric treatment as usual

SUMMARY:
Objective: This randomized and controlled trial was aimed at exploring the effect of a new mentalization-focused 4D interactive ultrasound and a week-by-week pregnancy diary intervention with substance-abusing pregnant women.

Method: Pregnant women referred to the hospital maternity outpatient clinic from primary health care due to substance abuse were recruited to participate in a randomized and controlled study. At admission, a psychiatric nurse offered all eligible women an opportunity for participation. A written informed consent was obtained from all participants included in the study. The participants were randomized into the intervention and control groups using a computer-generated block-randomization with block size of four. A separate randomization assignment was used for women in medication-assisted treatment for opioid dependence.

The intervention group subjects were offered three mentalization-focused interactive 4D ultrasounds at 24, 30 and 34 gestational weeks and a mentalization-focused week-by-week pregnancy diary combined with three antenatal sessions and an option for one diary session after delivery. The control group received active treatment as usual in an obstetric tertiary setting.

The pregnant woman and the child were followed-up until the child was one year old. The primary outcome was prenatal maternal depressive symptoms post-intervention, and secondary outcomes were anxiety symptoms, prenatal parental mentalization, maternal-fetal attachment and substance abuse. Other outcomes were utilisation of prenatal care, perinatal outcome, neonatal withdrawal symptoms and neonatal neurobehavior, postnatal maternal depressive and anxiety symptoms, parental mentalization, experienced stress from parenting and experienced social support, and emotional connection and commitment with the baby.

The study was conducted at the hospital maternity outpatient clinic for substance-abusing pregnant women at Turku University Hospital (Finland) between October 2011 and December 2015. The registration of the trial is made retrospectively, but the research plan and outcomes are reported in this registration as they were originally documented in the research plan approved by The Joint Ethics Committee of the University of Turku and the Hospital District of Southwest Finland on 14th of June 2011.

DETAILED DESCRIPTION:
Objective:

The aim of this controlled trial was to explore the effect of a new mentalization-focused 4D interactive ultrasound and a week-by-week pregnancy diary intervention with substance-abusing pregnant women.

Method:

This trial was conducted at the maternity outpatient clinic for substance-abusing pregnant women at Turku University Hospital, Finland, between October 2011 and December 2015. At Turku University Hospital there is a specialized antenatal outpatient clinic for pregnant women with substance abuse problems. Pregnant women referred to this facility from primary health care due to substance abuse were invited to participate the trial.

At admission, a psychiatric nurse offered all eligible women an opportunity to participate in the randomized trial. A written informed consent was obtained from all individual participants included in the study. The participants were randomized into the intervention and control groups using a computer-generated block-randomization with block size of four, and a separate randomization assignment was used for women in medication-assisted treatment for opioid addiction. In post-intervention phase at 35 gestational weeks, all participants were compensated with a 20 euros gift card targeted to the infant's needs. The research plan was approved by The Joint Ethics Committee of the University of Turku and the Hospital District of Southwest Finland on the 14th of June 2011.

Description of the intervention and the control condition:

The intervention group subjects were offered three mentalization-focused interactive 4D ultrasounds at 24, 30 and 34 gestational weeks and a mentalization-focused week-by-week pregnancy diary combined with three prenatal sessions and option for one diary session after delivery. Detailed intervention method description including a theoretical background of the intervention is already published and available (Pajulo et al. 2016).

1. Mentalization-focused interactive use of 4D ultrasound imaging:

   Three interactive 4D ultrasound sessions were offered for the intervention group participants at 24, 30 and 34 gestational weeks at the maternity outpatient clinic. The pregnant women participated in the sessions alone. The ultrasound sessions took around 20-30 minutes, and were performed by an experienced obstetrician and an infant mental health professional working in cooperation. The sessions were based on the intervention method called "ultrasound consultation" (Boukydis & Stockman, 2012; Boukydis, 2006) where the idea is to observe the fetus together with the parent(s); the fetal features, position, sleep-awake rhythm, personal characteristics, activities in the uterus and responses to mother's initiatives for interaction.The aim is to evoke the mother's active interest in this particular child and hence to enhance parental mentalization and maternal-fetal attachment.
2. The mentalization-focused week-by-week pregnancy diary:

To keep the fetus more actively in the mother's mind across pregnancy, a new mentalization-focused pregnancy diary was designed for the intervention group. Three prenatal meetings (45 minutes) with the infant mental health professional were offered for reflecting the mother's experiences on using the diary. The diary contains short sections for each pregnancy week including information about pregnancy, fetal development and health promoting practices. The key elements in the diary are the mentalization-focused questions and tasks encouraging the pregnant woman to reflect on her fetus and pregnancy and becoming a parent.

The control condition:

The intervention and control group received active treatment as usual in an obstetric tertiary setting, and treatment as usual formed the control condition for the intervention. The treatment was offered by a multidisciplinary team consisting of an obstetrician, a midwife, a social worker and a psychiatric nurse . The patients were referred to addiction and psychiatric treatment when needed. The Child Protection Services were involved in prenatal phase in accordance with the Finnish legislation.

Data collection:

The primary outcome was prenatal maternal depressive symptoms post-intervention, and secondary outcomes were anxiety symptoms, prenatal parental mentalization, maternal-fetal attachment and substance abuse. Other outcomes were utilisation of prenatal care, perinatal outcome, neonatal withdrawal symptoms and neonatal neurobehavior, postnatal maternal depressive and anxiety symptoms, parental mentalization, experienced stress from parenting and experienced social support, and emotional connection and commitment with the baby.

The pregnant woman and her child were followed-up until the child was one year old. The data was collected from multiple sources: standardized measures, questionnaires constructed for the study and information available from hospital medical records. As a part of routine clinical practice, the pregnant women were interviewed by the psychiatric nurse and the social worker. The interviews based on the European Addiction Severity Index-questionnaire (EuropASI) (Kokkevi & Hartgers, 1995), where the items regard maternal physical and mental health, substance abuse, employment and income, legal status and close relationships. Sociodemographic data was obtained by a ten-item questionnaire at baseline. Information regarding maternal psychiatric diagnosis and/or history was based on documented self-report or medical records. Information regarding maternal substance abuse was obtained through the medical records, and was based on maternal self-report or clinical documentation (intoxications, urine screening results, marks indicating intravenous substance abuse). Meconium sample was collected after birth for detection of illicit drugs. Data regarding utilisation of obstetric care and perinatal outcome was obtained from hospital medical records.

The standardized measures used to assess maternal depressive and anxiety symptoms, maternal-fetal attachment and parental mentalization were administered during pregnancy at two time points, i.e. before and after intervention (< 24th and > 34th gestational weeks, respectively). Routine postnatal follow-up visits at the socio pediatric unit were conducted when the infant was at 3 months and 1 year age. Standardized measures were administered during those follow-up visits to assess maternal postnatal depressive and anxiety symptoms, parental mentalization, experienced stress from parenting and experienced social support, and emotional connection and commitment with the baby. Medical records concerning health and psychosocial situation of the mother and infant were available, based on informed consent, until the child was one year old. The assessment time points and measures were the same for both groups.

The registration of the trial is made retrospectively, but the research plan and outcomes are reported in this registration as they were originally documented in the research plan approved by The Joint Ethics Committee of the University of Turku and the Hospital District of Southwest Finland on 14th of June 2011.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women referred to the hospital maternity outpatient clinic from primary health care due to substance abuse were recruited to participate in a randomized and controlled study. The subjects were referred from primary health care due to:

1. documented or self-reported illicit drug use, misuse of prescription medication or alcohol within three years prior to or during this pregnancy,
2. and/or sum score ≥ 3 points on TWEAK alcohol screening (Russell, 1994).

   The inclusion criteria included also:
3. pregnancy duration < 22 gestational weeks (gwks) at referral
4. singleton pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only pregnant women (pregnancy duration < 22 gestational weeks (gwks) at referral, and singleton pregnancy) were recruited
Enrollment: 126 (Actual)
Dates: Start 2011-10-18 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Prenatal depressive symptoms post-intervention at 35 gestational weeks | Post-intervention at 35 gestational weeks
  Assessment of prenatal depressive symptoms with Edinburgh Pre/Postnatal Depression Scale (EPDS); theoretical range of total scale (minimum and maximum scores) 0-30 points and lower total score indicating lower level of depressive symptoms and better outcome.

SECONDARY OUTCOMES:
Prenatal parental mentalization post-intervention at 35 gestational weeks | Post-intervention at 35 gestational weeks
  Assessment of prenatal parental mentalization with Prenatal Parental Reflective Functioning Questionnaire (P-PRFQ): theoretical range of the sum index is 1-7 points (minimum and maximum scores), and higher total score is indicating higher level of parental mentalization and better outcome.
Maternal-fetal attachment post-intervention at 35 gestational weeks | Post-intervention at 35 gestational weeks
  Assessment of maternal-fetal attachment with Maternal-fetal Attachment Scale (MFAS): theoretical range of total scale is 24-120 points (minimum and maximum scores), and higher total score is indicating stronger maternal-fetal attachment and better outcome.
Prenatal maternal substance abuse (health behaviour) | From date of randomization until the date of delivery, assessed up to 42 gestational weeks
  Prenatal clinical assessments of prenatal substance abuse documented in the hospital medical records (intoxications, urine screening results, marks indicating intravenous substance abuse): The more findings, the worse the outcome.
Prenatal anxiety symptoms post-intervention at 35 gestational weeks | Post-intervention at 35 gestational weeks
  Assessment of prenatal anxiety symptoms with The State Section of The State-Trait Anxiety Inventory (STAI): theoretical range of total scale is 20-80points (minimum and maximum scores), and lower total score is indicating lower level of prenatal anxiety and better outcome.

OTHER OUTCOMES:
Prenatal care | From date of randomization until the date of delivery, assessed up to 42 gestational weeks
  Utilization of obstetric and emergency department hospital care at the Turku University Hospital (medical record data concerning outpatient visits, hospital admissions)
Neonatal child outcome: Birth weight | After birth up to 1 day
  Birth weight of the neonate in grams(g)
Neonatal child outcome: Gestational age | After birth up to 1 day
  Gestational age of the neonate in gestational weeks
Neonatal child outcome: Apgar Score at 5 minutes | 5 minutes after birth
  Apgar score of the neonate at 5 minutes age. Apgar score total range is 0-10 points (minimum and maximum scores), and higher total score indicates better neonatal outcome
Neonatal child outcome: Head circumference | After birth up to 1 day
  Head circumference in centimeters(cm)
Neonatal child outcome: Length of hospital stay after birth | After birth up to 1 month
  Duration of the neonate's hospital care in days
Fetal drug exposure | After birth up to 7 days
  Meconium sample for testing exposure to illicit drugs
Postnatal depressive symptoms | 3 months and 1 year after delivery
  Assessment of postnatal depressive symptoms with Edinburgh Postnatal Depression Scale (EPDS); theoretical range of the total scale is 0-30 points (minimum and maximum scores), and lower total score is indicating lower level of depressive symptoms and better outcome.
Postnatal anxiety symptoms | 3 months and 1 year after delivery
  Assessment of postnatal anxiety symptoms with The State Section of The State-Trait Anxiety Inventory (STAI): theoretical range of the total scale is 20-80 points (minimum and maximum scores), and lower total score is indicating lower level of postnatal anxiety and better outcome.
Postnatal parental mentalization | 3 months and 1 year after delivery
  Assessment of postnatal parental mentalization with Parental Reflective Functioning Questionnaire (PRFQ): theoretical range sum index 1-7 points, higher score indicating better outcome (higher mentalization)
Experienced parenting stress and social support | 3 months and 1 year after delivery
  Assessment of experienced stress in parenting and social support with Parenting Stress Index and Social Support (SPSQ): 15 items in section measuring experienced stress, sum index theoretical range 1-5 points (minimum and maximum scores), higher score indicating worse outcome (higher stress).
Emotional connection and commitment with the baby | 3 months and 1 year after delivery
  Assessment of mother's emotional connection and commitment with the baby with Postpartum Bonding Questionnaire (PBQ): theoretical range sum index 1-5 (minimum and maximum scores), higher score indicating worse outcome (weaker bonding)
Neonatal neurobehavior status | After birth up to 7 days
  Assessment of neonatal neurobehavior with Dubowitz Scale: 34 items scored with theoretical range 0-1 and total score theoretical range 0-34 points (minimum and maximum scores), higher score indicating better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Eeva Ekholm, MD, PhD, Principal Investigator — Department of Obstetrics and Gynecology, Turku University Hospital, Kiinamyllynkatu 4-8, PL 52, 20521 Turku, Finland Department of Obstetrics and Gynecology, University of Turku, 20014 Turku, Finland; Marjukka Pajulo, MD, PhD, Principal Investigator — Department of Child Psychiatry, Turku University Hospital, Kiinamyllynkatu 4-8, PL 52, 20521 Turku, Finland Department of Child Psychiatry and Finn Brain, University of Turku, 20014 Turku, Finland
Locations (1):
- Department of Obstetrics and Gynecology and Department of Child Psychiatry, Turku University Hospital; Department of Obstetrics and Gynecology and Department of Child Psychiatry, University of Turku, Turku, Finland, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boukydis CF, Treadwell MC, Delaney-Black V, Boyes K, King M, Robinson T, Sokol R. Women's responses to ultrasound examinations during routine screens in an obstetric clinic. J Ultrasound Med. 2006 Jun;25(6):721-8. doi: 10.7863/jum.2006.25.6.721. PMID 16731888
- [Background] Boukydis Z. Ultrasound consultation to reduce risk and increase resilience in pregnancy. Ann N Y Acad Sci. 2006 Dec;1094:268-71. doi: 10.1196/annals.1376.032. PMID 17347359
- [Background] Kokkevi, A., & Hartgers, C. (1995). EuropASI: European adaptation of a multidimensional assessment instrument for drug and alcohol dependence. Eur Addict Res, 1, 208-210.
- [Background] Pajulo H, Pajulo M, Jussila H, Ekholm E. SUBSTANCE-ABUSING PREGNANT WOMEN: PRENATAL INTERVENTION USING ULTRASOUND CONSULTATION AND MENTALIZATION TO ENHANCE THE MOTHER-CHILD RELATIONSHIP AND REDUCE SUBSTANCE USE. Infant Ment Health J. 2016 Jul;37(4):317-34. doi: 10.1002/imhj.21574. Epub 2016 Jun 24. PMID 27341555
- [Background] Russell M. New Assessment Tools for Risk Drinking During Pregnancy: T-ACE, TWEAK, and Others. Alcohol Health Res World. 1994;18(1):55-61. PMID 31798157
- [Derived] Jussila H, Pajulo M, Ekholm E. A Novel 4D Ultrasound Parenting Intervention for Substance Using Pregnant Women in Finland: Participation in Obstetric Care, Fetal Drug Exposure, and Perinatal Outcomes in a Randomized Controlled Trial. Matern Child Health J. 2020 Jan;24(1):90-100. doi: 10.1007/s10995-019-02773-w. PMID 31250239